CLINICAL TRIAL: NCT03292965
Title: Monitoring of Postoperative Residual Neuromuscular Blockade in Laparoscopic Surgery: Comparison of Neostigmine and Sugammadex
Brief Title: Monitoring of Postoperative Residual Neuromuscular Blockade in Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, LEE YEA JI, clinical professor of department of anesthesiology and pain medicine, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: B-1609-363-002
Record Dates: First submitted 2017-09-21; First posted 2017-09-26 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Neuromuscular Block, Residual
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Neostigmine; Sugammadex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neostigmine (Active Comparator): At the end of surgery, administrating neostigmine to participants according to the protocol below:
  when train-of-four (TOF) 2-3, administrating neostigmine 50mcg/kg when TOF 4 with fade, administrating neostigmine 40mcg/kg when TOF 4 without fade, administrating neostigmine 20mcg/kg
  Interventions: Drug: Neostigmine
- Sugammadex (Active Comparator): At the end of surgery, administrating sugammadex to participants according to the protocol below:
  when TOF=0 and post-tetanic count (PTC)=1 or more, administrating sugammadex 4mg/kg when TOF=1 or more, administrating sugammadex 2mg/kg when TOF 4 without fade, administrating neostigmine 20mcg/kg
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Neostigmine — Referring to the randomisation allocation program, participants allocated to group neostigmine, administrate neostigmine as reversal
  Arms: Neostigmine
Drug: Sugammadex — Referring to the randomisation allocation program, participants allocated to group sugammadex, administrate sugammadex as reversal
  Other Names: Bridion
  Arms: Sugammadex

SUMMARY:
Compare the reversal effect of neostigmine and sugammadex using quantitative neuromuscular monitoring

DETAILED DESCRIPTION:
At the end of surgery, decide the dosage of reversal referring to quantitative neuromuscular monitoring value (TOF). After the administration of reversal, the anesthesiologist who are going to manage the participant should not check the quantitative neuromuscular monitoring and determine the timing of extubation only with his (or her) judgement. After entering post-anaesthesia care unit (PACU) measure the TOF value and check the incidence of TOF ratio > 0.9 between the neostigmine group and sugammadex group.

ELIGIBILITY:
Inclusion Criteria:

* patients aged over 18 years, planned to undergoing elective laparoscopic surgery under general anesthesia

Exclusion Criteria:

* Obesity BMI over 30 kg/m2
* Impairment of renal or/and liver function
* Allergy to rocuronium, sugammadex
* (Familial) history of malignant hyperthermia
* Taking medicines which is affecting neuromuscular function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
the incidence of postoperative residual curarization | Immediately after entering PACU
  definition of postoperative residual curarization: TOF ration is 0.9 or over 0.9

CONTACTS AND LOCATIONS:
Overall Officials: AhYoung Oh, M.D Ph. D, Study Chair — Department of anesthesiology and pain medicine
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee YJ, Oh AY, Koo BW, Han JW, Park JH, Hong JP, Seo KS. Postoperative residual neuromuscular blockade after reversal based on a qualitative peripheral nerve stimulator response: A randomised controlled trial. Eur J Anaesthesiol. 2020 Mar;37(3):196-202. doi: 10.1097/EJA.0000000000001157. PMID 31977627